CLINICAL TRIAL: NCT03059082
Title: A Critical Illness Recovery Navigator for Alcohol: a Pilot Clinical Trial
Brief Title: A Critical Illness Recovery Navigator for Alcohol
Acronym: CIRNA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator surrendered funding and left institution.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 16-2094
Record Dates: First submitted 2017-01-03; First posted 2017-02-23 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continued Interaction (Other): This group will undergo contact with Recovery Navigator on an "as needed basis" up to 6 months.They will then have a 3 month and 6 month follow up visit with the PI. There is no drug or treatment administered to the subject. The intervention is the conversation/contact with the Recovery Navigator, in this arm, it is continued throughout the study.
  Note: The first 10 subjects will not be randomized and will be assigned to this Arm. The purpose of this is to ensure the fidelity of the intervention. The remaining 60 subjects will be randomized equally among the three Arms. Data from the first 10 subjects will not be considered for the outcome measures.
  Interventions: Behavioral: Recovery Navigator on an as needed basis up to 6 months
- Single interaction (Other): This group will undergo one interaction with the Recovery Navigator prior to the hospital discharge. They will then have a 3 month and 6 month follow up visit with the PI. There is no drug or treatment administered to the subject.The intervention is the conversation/contact with the Recovery Navigator, in this arm, it is conducted once.
  Interventions: Behavioral: Recovery Navigator prior to hospital discharge
- Control (Other): This group will not have any interaction with the Recovery Navigator. They will then have a 3 month and 6 month follow up visit. There is no drug or treatment administered to the subject.
  Interventions: Other: No interaction with Recovery Navigator

INTERVENTIONS:
Behavioral: Recovery Navigator on an as needed basis up to 6 months — This group will undergo contact with Recovery Navigator on an "as needed basis" up to 6 months and then have a 3 month and 6 month follow-up visit.
  Other Names: Recovery Navigator
  Arms: Continued Interaction
Behavioral: Recovery Navigator prior to hospital discharge — This group will undergo one interaction with Recovery Navigator prior to hospital discharge and then have a 3 month and 6 month follow-up visit.
  Other Names: Recovery Navigator
  Arms: Single interaction
Other: No interaction with Recovery Navigator — This group will not have any interaction with Recovery Navigator. They will have a 3 month and 6 month follow-up visit.
  Other Names: Control
  Arms: Control

SUMMARY:
Excessive alcohol consumption is common in patients admitted to the intensive care unit (ICU). Among patients who survive an ICU admission, excessive alcohol consumption is associated with a higher risk of being admitted the hospital. In this study, the Investigators will compare an intervention designed to address excessive drinking in ICU survivors to usual care. This intervention combines motivational interviewing (MI) and shared decision making (SDM). MI and SDM share several core components including the development of a therapeutic alliance and promotion of autonomy. MI can be employed in the context of motivating a patient to change their drinking. Once this decision has been made, SDM can be employed to help a patient decide amongst multiple reasonable treatment options. The Investigators long-term goal is to test whether MI-SDM is better than usual care and whether multiple sessions of MI-SDM are better than a single session. This pilot clinical trial will demonstrate the feasibility of conducting a larger efficacy study to test these hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to the intensive care unit;
2. Age 18 years or older;
3. Resolution of critical illness, defined as the intention of the treating team to discharge the patient or downgrade their admission level from the ICU to a progressive care unit or the floor;
4. Resolution of delirium, defined by:

   * a Riker Agitation Sedation Scale score of 0,
   * a negative CAM ICU, and
   * confirmation from the treating team (nurse, physicians) that the patient is not delirious.
5. AUDIT-C score of 3 or greater for women and 4 or greater for men.

Exclusion Criteria:

1. Prisoner;
2. Pregnant;
3. Unable to speak or write in English;
4. Unable to provide informed consent;
5. Unable to provide a home or cell phone number plus at least one additional way to be contacted (mail, email, friend or family);
6. Expected survival less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-12; Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction and Acceptability of study | 6 months
  Client satisfaction questionnaire (CSQ-8), with revisions to make it specific to the objectives of this study.

SECONDARY OUTCOMES:
Subject Recruitment Rate | 6 months
  The following will be collected to determine the feasibility and design of a larger effectiveness study: recruitment rates calculated as the number of patients recruited per month per hospital.
Subject willingness to be randomized | 6 months
  The number of patients who refuse study participation due to refusal to undergo randomization. This will be collected to inform the feasibility and design of a larger effectiveness study.
Subject Dropout Rates | 3 and 6 months
  The percentage of subjects who do not show up for study visits calculated for each arm of the study.
Subjects with at least one visit after discharge | 6 months
  The percentage of subjects with at least one visit after discharge with the navigator.
Time per subject visit | 6 months
  The amount of time per subject visit to determine feasibility of the intervention for a larger study.
Number of visits | 6 months.
  the Number of visits total to help determine feasibility of the intervention for a larger study.
Initiation of treatment within 14 days. | 14 days
  Initiation of treatment by attendance at one treatment session within 14 days as efficacy measure for larger trial.
Initiation of alcohol/drug treatment within 6 months | 6 months
  Initiation of treatment by attendance at one treatment session within 6 months as efficacy measure for larger trial
Engagement in alcohol/drug treatment | 3 and 6 months
  2 or more inpatient admissions, outpatient visits, intensive outpatient encounters or partial hospitalizations as efficacy measure for larger trial
Completion of alcohol/drug treatment | 3 and 6 months
  Completion of alcohol treatment program as efficacy measure for larger trial
Hospital re admissions and emergency department visits | 3 and 6 months
  Number of hospital readmission and emergency department visits as efficacy measure for larger trial
Receipt of treatment for drug problems | 3 and 6 months
  Receipt of treatment for drug problems as efficacy measure for larger trial.
Receipt of psychiatric treatment. | 3 and 6 months
  Receipt of psychiatric treatment as efficacy measure for larger trial.
Number of days abstained from alcohol consumption | 30 days
  Percentage of days abstinent from alcohol consumption in 30 day timeframe
Number of days with reported heavy alcohol consumption | 30 days
  Percentage of days with reported heavy alcohol consumption in 30 day timeframe
Phosphatidylethanol (PEth) level at 6 months | 6 months
  Phosphatidylethanol (PEth) level at 6 months compared against subject's self-reported alcohol consumption and measured by United States Drug Testing laboratory
Alcohol related problems measured by SIP-2R | 3 and 6 months
  alcohol related problems assessed by administering the Short Inventory of Problems 2, revised (SIP-2R).
HADS anxiety assessment | 3 and 6 months
  Anxiety assessed with 14 item Hospital Anxiety and Depression Scale (HADS).
HADS depression assessment | 3 and 6 months
  Depression assessed with 14 item Hospital Anxiety and Depression Scale (HADS).
Post Traumatic Stress Disorder (PTSD) symptoms | 3 and 6 months.
  PTSD symptoms assessed using the Impact of Events Scale, revised.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan J Clark, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States